CLINICAL TRIAL: NCT04750174
Title: Effectiveness of Kinesiotape on Children With Cerebral Palsy and Oropharyngeal Dysphagia
Brief Title: Kinesiotape and Dysphagia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Gaziantep (Other)
Responsible Party: Principal Investigator, Mazlum Serdar Akaltun, Assistant Professor, University of Gaziantep
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MSAkaltun
Record Dates: First submitted 2021-02-06; First posted 2021-02-11 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Dysphagia; Cerebral Palsy
Keywords: Kinesiotape; Swallowing; Cerebral Palsy; Dysphagia
MeSH Terms: conditions — Deglutition Disorders; Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Patients who met the study criteria were assigned to either the intervention group or the sham group after being questioned to provide their caregivers understanding of all study procedures and requirements for participation.
Who Masked: Participant, Investigator
Masking Description: A short practical training was performed before the study. The study was performed by a group of independent specialists blinded to treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesiotape Group (Active Comparator): In active group, KT was applied with stretching to the suprahyoid muscles with right method.
  Interventions: Other: Kinesiotaping
- Sham Kinesiotape Group (Sham Comparator): In sham group, KT was applied without stretching to the suprahyoid region and not including the origins of mylohyoid and digastric muscles
  Interventions: Other: Kinesiotaping

INTERVENTIONS:
Other: Kinesiotaping — Kinesiotape (KT) has been used by Dr. Kenzo Kase for the first time as based on the opinion that more successful results can be obtained in a banding method similar to the structural characteristics and flexibility of human skin without limiting the joint movements for edema control, joint protection, and proprioception training. In recent years, KT have been applied with a wide variety of techniques including muscle techniques for the inhibition and stimulation of muscles, fascia correction technique which aims to reduce tension and adhesions by making vibration movement between the fascia layers and field correction technique aiming to reduce regional pressure in the presence of pain, inflammation or edema as well as lymphatic correction technique for regulating lymphatic circulation .

SUMMARY:
Dysphagia is common problem in almost all children with cerebral palsy (CP) and there is no consensus about to dysphagia therapy modalities.We aimed to investigate the short- and long-term effects of kinesio taping (KT) on dysphagia in children with CP.

DETAILED DESCRIPTION:
There is a few studies for the effectiveness of KT application in the treatment of dysphagia and its effectiveness is controversial. These small-scale studies conducted to improve control of drooling in the oral phase of swallowing in CP. However, there are no studies that have evaluated swallowing as a whole. Moreover, there is a need to carry out studies evaluating the efficacy of KT in dysphagia treatment with a high level of evidence and duration of effectivenes for a period longer than 3 months. This study is designed to answer the following research questions: "Is KT application effective in the treatment of dysphagia in CP?" ''If it is effective, whether the effect of KT therapy persists more than 3 months''.

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of 2 and 6 years who had oropharyngeal dysphagia (OD) symptom and/or finding and were subsequently hospitalized and rehabilitated were included in this study.

Exclusion Criteria:

* Patients with history of maxillary, head or neck surgery or botulinum toxin injection, structural oropharyngeal abnormality, known esophageal dysphagia and/or gastroesophageal reflux disease, who were received medical and/or physical therapy for dysphagia in the last 6 months, using drugs for seizures or spasticity as well as no oral intake and tube dependent completely for feeding were not included.

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Functional oral intake scale | 6th week
  The scale evaluates the patient's safe and adequate functional oral intake and consists of 7 levels.

SECONDARY OUTCOMES:
Family satisfaction level | 18th week
  Children's primary caregivers were asked to evaluate the change in swallowing of children at 6th and 18th weeks with 5-point Likert scale. Accordingly, "so much better" to "so much worse" were scored between 1 and 5.

CONTACTS AND LOCATIONS:
Overall Officials: Mazlum Serdar Akaltun, M.D., Principal Investigator — University of Gaziantep
Locations (1):
- Gaziantep University, Gaziantep, Turkey (Türkiye)